CLINICAL TRIAL: NCT01714505
Title: Early Feasibility Study 2 of Outpatient Control-to-Range - Testing System Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Sansum Diabetes Research Institute (Other); University of Padova (Other); University Hospital, Montpellier (Other)
Responsible Party: Principal Investigator, Boris Kovatchev, PhD, Director, UVA Center for Diabetes Technology, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16457; JDRF 22-2011-649 (Other Grant/Funding Number: Juvenile Diabetes Research Foundation)
Record Dates: First submitted 2012-10-23; First posted 2012-10-26 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Continuous Glucose Monitor; Artificial Pancreas; Insulin Pump; Closed Loop control; Open Loop treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Involving Automated CTR (Experimental): Closed-Loop Control: Insulin delivery will be controlled by the Diabetes Assistant (DiAs) system running in Control to Range (CTR) or in Safety Only mode. The subject will interact with the system through its Graphic User Interface (GUI). Subjects will not be allowed to administer correction boluses between meals and snacks as the DiAs will automatically be adjusting insulin to correct for hyperglycemia. The total doses recommended by the DiAs prior to meals and snacks includes the correction dose and Insulin on Board (IOB) calculated by the system.
  Interventions: Device: Diabetes Assistant (DiAs)
- CGM-Augmented Insulin Pump Treatment (No Intervention): Open Loop Control: Insulin delivery will be controlled by the Diabetes Assistant (DiAs) system running in open-loop mode. The subject will interact with the system through its Graphic User Interface (GUI). Subjects will be permitted to administer correction boluses at any time during the Control Admission, whether or not they are eating a scheduled meal or snack. DiAs will be initialized with the subject's typical insulin pump settings. The subject will be reminded that all treatment decisions should be based on fingerstick values and not on continuous glucose monitor (CGM) values.

INTERVENTIONS:
Device: Diabetes Assistant (DiAs) — A medical platform that uses a smart-phone to connect to a continuous glucose sensor to insulin pump and run closed-loop control. The cell phone runs the Control to Range and is connected to work with the insulin pump and continuous glucose monitor to help keep the blood sugar in a desired range (80-180 mg/dL during the day) and help avoid hypoglycemia during the night.
  Arms: Experimental Involving Automated CTR

SUMMARY:
An unblinded, randomized, cross-over design with each patient participating in two 40-hour outpatient admissions: (a) Experimental involving automated Control-to-Range (CTR) and (b) Control using Continuous Glucose Monitor (CGM)- augmented insulin pump treatment outside of a hospital based clinical research center. The principal goal is to validate a smart phone-based control-to-range (CTR) system for ambulatory use and to estimate the effect of CTR vs. sensor-augmented pump therapy, thereby providing justification for further larger home-based trials of CTR.

DETAILED DESCRIPTION:
The overall objective of this project is to sequentially test, validate, obtain regulatory approval for, and deploy at home, a closed-loop Control-to-Range (CTR) system for optimal blood glucose (BG) regulation in people with type 1 diabetes. The CTR system is comprised of two algorithmic layers: a Safety Supervision Module (SSM) and Insulin on Board Tracking and Safety Module (ITSM), and an automated Range Correction Module (RCM). Both modules will receive continuous glucose monitoring (CGM) and insulin delivery data. The SSM and ITSM will monitor the safety of the subject's continuous subcutaneous insulin infusion pump (CSII) to prevent hypoglycemia. The RCM will be responsible for optimizing BG control and mitigating postprandial hyperglycemic excursions through series of insulin boluses. To run CTR, we will use our wearable artificial pancreas platform, known as DiAs (Diabetes Assistant), which consists of a smart phone running CTR and connected to standard insulin delivery and CGM devices.

ELIGIBILITY:
Inclusion Criteria:

1. ≥21 and <65 years old.
2. Clinical diagnosis of type 1 diabetes mellitus. For an individual to be enrolled at least one criterion from each list must be met.

   o Criteria for documented hyperglycemia (at least 1 must be met): i. Fasting glucose ≥126 mg/dL - confirmed ii. Two-hour Oral Glucose Tolerance Test (OGTT) glucose ≥200 mg/dL - confirmed iii. HbA1c ≥6.5% documented - confirmed iv. Random glucose ≥200 mg/dL with symptoms v. No data at diagnosis is available but the participant has a convincing history of hyperglycemia consistent with diabetes

   o Criteria for requiring insulin at diagnosis (1 must be met): i. Participant required insulin at diagnosis and continually thereafter ii. Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did require insulin eventually and used continually iii. Participant did not start insulin at diagnosis but continued to be hyperglycemic, had positive islet cell antibodies - consistent with latent autoimmune diabetes in adults (LADA) and did require insulin eventually and used continually
3. Use of an insulin pump to treat his/her diabetes for at least 1 year.
4. Familiarity with a bolus calculator with the current insulin pump with pre-defined parameters for carbohydrate (CHO) ratio, insulin sensitivity factor (ISF), target glucose and active insulin.
5. HbA1c <9% as measured with DCA2000 or equivalent device.
6. Not currently known to be pregnant, breast feeding, or intending to become pregnant (females).
7. Demonstration of proper mental status and cognition for the study.
8. Willingness to avoid consumption of acetaminophen-containing products during the study interventions involving CGM use.
9. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, have stability on the medication for at least 2 months prior to enrollment in the study.

Exclusion Criteria:

1. Severe hypoglycemia resulting in seizure, loss of consciousness, or diabetic ketoacidosis within the 12 months prior to enrollment.
2. Pregnancy; breast feeding, or intention of becoming pregnant.
3. Uncontrolled arterial hypertension (Resting diastolic blood pressure >90 mmHg and/or systolic blood pressure >160 mmHg).
4. Conditions which may increase the risks associated with possible hypoglycemia, such as any active cardiac disorder/arrhythmia, uncontrolled coronary artery disease during the previous year (e.g. history of myocardial infarction, acute coronary syndrome, therapeutic coronary intervention, coronary bypass or stenting procedure, stable or unstable angina, episode of chest pain of cardiac etiology with documented EKG changes, or positive stress test or catheterization with coronary blockages >50%), congestive heart failure, history of cerebrovascular event, seizure disorder, syncope, adrenal insufficiency, neurologic disease or atrial fibrillation.
5. Self-reported hypoglycemia unawareness.
6. History of a systemic or deep tissue infection with methicillin-resistant staph aureus or Candida albicans.
7. Use of a device that may pose electromagnetic compatibility issues and/or radiofrequency interference with the CGM (implantable cardioverter-defibrillator, electronic pacemaker, neurostimulator, intrathecal pump, and cochlear implants).
8. Anticoagulant therapy other than aspirin.
9. Oral steroids.
10. Medical condition requiring use of an acetaminophen-containing medication that cannot be withheld for the study admissions.
11. Psychiatric disorders that would interfere with study tasks (e.g. inpatient psychiatric treatment within 6 months prior to enrollment).
12. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
13. Known current or recent alcohol or drug abuse.
14. Medical conditions that would make operating a CGM, the DiAs cell phone or insulin pump difficult (e.g. blindness, severe arthritis, immobility).
15. Any skin condition that prevents sensor or pump placement on the abdomen or arm (e.g. bad sunburn, pre-existing dermatitis, intertrigo, psoriasis, extensive scarring, cellulitis).
16. In adherence with the One Touch Ultra 2 User Guide, subjects with hematocrit levels less than 30% and above 55% will be excluded.
17. Impaired hepatic function measured as alanine aminotransferase or aspartate aminotransferase ≥three times the upper reference limit.
18. Impaired renal function measured as creatinine >1.2 times above the upper limit of normal.
19. Uncontrolled microvascular (diabetic) complications, such as current proliferative diabetic retinopathy or macular edema, known diabetic nephropathy (other than microalbuminuria with normal creatinine) or neuropathy requiring treatment.
20. Active gastroparesis requiring current medical therapy.
21. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study.
22. Uncontrolled thyroid disease.
23. Known bleeding diathesis or dyscrasia.
24. Known allergy to medical adhesives, components of the insulin pump insertion set or continuous glucose monitor sensor.
25. Active enrollment in another clinical trial.
26. Use of anti-diabetic agents other than continuous subcutaneous insulin infusion (CSII) including long-acting insulin, intermediate-acting insulin, metformin, sulfonylureas, meglitinides, thiazolidinediones, DPP-IV inhibitors, glucagon-like peptide 1 agonists, and alpha-glucosidase inhibitors
27. Subjects with basal rates less than 0.01U/hr.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris P. Kovatchev, Ph.D., Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Result] Kovatchev BP, Renard E, Cobelli C, Zisser HC, Keith-Hynes P, Anderson SM, Brown SA, Chernavvsky DR, Breton MD, Mize LB, Farret A, Place J, Bruttomesso D, Del Favero S, Boscari F, Galasso S, Avogaro A, Magni L, Di Palma F, Toffanin C, Messori M, Dassau E, Doyle FJ 3rd. Safety of outpatient closed-loop control: first randomized crossover trials of a wearable artificial pancreas. Diabetes Care. 2014 Jul;37(7):1789-96. doi: 10.2337/dc13-2076. Epub 2014 Jun 14. PMID 24929429

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-Loop Then Closed-Loop Control: Open-Loop: Insulin delivery will be controlled by the DiAs system running in open-loop mode. The subject will interact with the system through its GUI. Subjects will be permitted to administer correction boluses at any time during the Control Admission, whether or not they are eating a scheduled meal or snack. DiAs will be initialized with the subject's typical insulin pump settings.
  Closed-Loop: Insulin delivery will be controlled by the Diabetes Assistant (DiAs) system running in Control to Range (CTR) or in Safety Only mode. The subject will interact with the system through its Graphic User Interface (GUI). Subjects will not be allowed to administer correction boluses between meals and snacks as the DiAs will automatically be adjusting insulin to correct for hyperglycemia.
- Closed-Loop Then Open-Loop Control: Closed-Loop: Insulin delivery will be controlled by the Diabetes Assistant (DiAs) system running in Control to Range (CTR) or in Safety Only mode. The subject will interact with the system through its Graphic User Interface (GUI). Subjects will not be allowed to administer correction boluses between meals and snacks as the DiAs will automatically be adjusting insulin to correct for hyperglycemia.
  Open-Loop: Insulin delivery will be controlled by the DiAs system running in open-loop mode. The subject will interact with the system through its GUI. Subjects will be permitted to administer correction boluses at any time during the Control Admission, whether or not they are eating a scheduled meal or snack. DiAs will be initialized with the subject's typical insulin pump settings.
Period: Admission 1 (40 Hours)
Arm/Group | Open-Loop Then Closed-Loop Control | Closed-Loop Then Open-Loop Control
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Period: Admission 2 (40 Hours)
Arm/Group | Open-Loop Then Closed-Loop Control | Closed-Loop Then Open-Loop Control
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Open and Closed Loop Control: Closed-Loop: Insulin delivery will be controlled by the Diabetes Assistant (DiAs) system running in Control to Range (CTR) or in Safety Only mode. The subject will interact with the system through its Graphic User Interface (GUI). Subjects will not be allowed to administer correction boluses between meals and snacks as the DiAs will automatically be adjusting insulin to correct for hyperglycemia.
  Open-Loop: Insulin delivery will be controlled by the DiAs system running in open-loop mode. The subject will interact with the system through its GUI. Subjects will be permitted to administer correction boluses at any time during the Control Admission, whether or not they are eating a scheduled meal or snack. DiAs will be initialized with the subject's typical insulin pump settings.
Arm/Group | Open and Closed Loop Control
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Safety, Low Blood Glucose Index (LBGI)
Description: The LBGI reflects the frequency and extent of hypoglycemic episodes and presents the results in "risk space." Thus the LBGI is a weighted average of the number of hypoglycemic readings, with progressively increasing weights as BG levels go down. The increase of the weights follows a risk function; thus the LBGI has been associated with risk for hypoglycemia and prediction of severe hypoglycemic episodes.
  LBGI < 2.5 is associated with low risk of hypoglycemia, 2.5 < LBGI < 5 is associated with a moderate risk of hypoglycemia and LBGI > 5 is associated with a high risk of hypoglycemia.
Time Frame: 40 hours (x2 admissions)
Measure: Mean (Standard Deviation); unit: index score
Groups:
- Closed-loop Control to Range: Closed-Loop Control: Insulin delivery will be controlled by the Diabetes Assistant (DiAs) system running in Control to Range (CTR) or in Safety Only mode. The subject will interact with the system through its Graphic User Interface (GUI). Subjects will not be allowed to administer correction boluses between meals and snacks as the DiAs will automatically be adjusting insulin to correct for hyperglycemia. The total doses recommended by the DiAs prior to meals and snacks includes the correction dose and Insulin on Board (IOB) calculated by the system.
  Diabetes Assistant (DiAs): A medical platform that uses a smart-phone to connect to a continuous glucose sensor to insulin pump and run closed-loop control. The cell phone runs the Control to Range and is connected to work with the insulin pump and continuous glucose monitor to help keep the blood sugar in a desired range (80-180 mg/dL during the day) and help avoid hypoglycemia during the night.
- Open-Loop CGM-Augmented Insulin Pump Therapy: Open Loop Control: Insulin delivery will be controlled by the Diabetes Assistant (DiAs) system running in open-loop mode. The subject will interact with the system through its Graphic User Interface (GUI). Subjects will be permitted to administer correction boluses at any time during the Control Admission, whether or not they are eating a scheduled meal or snack. DiAs will be initialized with the subject's typical insulin pump settings. The subject will be reminded that all treatment decisions should be based on fingerstick values and not on continuous glucose monitor (CGM) values.
Arm/Group | Closed-loop Control to Range | Open-Loop CGM-Augmented Insulin Pump Therapy
Number analyzed (Participants) | 18 | 18
index score | 0.64 (0.72) | 1.12 (0.77)
Statistical Analysis 1: Comparison: Closed-loop Control to Range vs Open-Loop CGM-Augmented Insulin Pump Therapy; Test type: Superiority or Other; p = 0.003, t-test, 1 sided; Paired t-tests: compare LBGI, carbohydrates for hypoglycemia treatment, % of time in range and average BG on CLC vs OL

2. Secondary Outcome: Efficacy, Time Spent in Target Range
Description: Percentage of time in the target range of 3.9-10 mmol/L (70-180 mg/dL).
Time Frame: 40 hours (x2 admissions)
Measure: Mean (Standard Deviation); unit: percentage of time spent in range
Arm/Group | Closed-loop Control to Range | Open-Loop CGM-Augmented Insulin Pump Therapy
Number analyzed (Participants) | 18 | 18
percentage of time spent in range | 66.1 (18.6) | 70.7 (21.7)
Statistical Analysis 1: Comparison: Closed-loop Control to Range vs Open-Loop CGM-Augmented Insulin Pump Therapy; Test type: Superiority or Other; p > 0.1, t-test, 1 sided

3. Primary Outcome: Safety, Frequency of Hypoglycemia
Description: Hypoglycemic episodes are defined as BG < 3.9mmol/L
Time Frame: 40 hours (x 2 admissions)
Measure: Mean (Standard Deviation); unit: hypoglycemic episodes/participant
Arm/Group | Closed-loop Control to Range | Open-Loop CGM-Augmented Insulin Pump Therapy
Number analyzed (Participants) | 18 | 18
hypoglycemic episodes/participant | 1.22 (0.4) | 2.39 (0.6)
Statistical Analysis 1: Comparison: Closed-loop Control to Range vs Open-Loop CGM-Augmented Insulin Pump Therapy; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Closed-loop Control to Range | Open-Loop CGM-Augmented Insulin Pump Therapy
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 5/19 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closed-loop Control to Range (N=19) | Open-Loop CGM-Augmented Insulin Pump Therapy (N=20)
Hyperglycemia (Endocrine disorders) | 3 (3) | 0 (0)
System Malfunction (Investigations) | 2 (2) | 0 (0)
Hyper and Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1) — Patient was referred to endocrinologist for inappropriate pump parameters.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes